CLINICAL TRIAL: NCT04938687
Title: Pilot, Effect of Respiratory-Gated Auricular Vagal Afferent Nerve Stimulation (RAVANS) on Post-Treatment Lyme Disease Syndrome
Brief Title: Effect of Auricular Vagal Nerve Electrical Stimulation on Post-Treatment Lyme Disease Syndrome
Acronym: RavLyme
Status: Completed | Type: Interventional
Sponsor: Spaulding Rehabilitation Hospital (Other)
Responsible Party: Principal Investigator, Qing Mei Wang, M.D., Director, Stroke Biological Recovery Laboratory, Spaulding Rehabilitation Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2021P000566
Record Dates: First submitted 2021-06-09; First posted 2021-06-24 (Actual); Results first posted 2025-11-10 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2025-09

CONDITIONS: Post-Treatment Lyme Disease Syndrome
MeSH Terms: conditions — Post-Lyme Disease Syndrome

STUDY DESIGN:
Intervention Model Description: randomized, double blinded, sham-controlled
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | Unapproved Device: Yes

ARMS (2):
- RAVANS (Experimental): active RAVANS, 20 minutes each treatment, 3 times per week for 2 weeks
  Interventions: Device: respiratory-gated auricular vagal afferent nerve stimulation (RAVANS)
- Sham stimulation (Sham Comparator): Sham-stimulation, 20 minutes each treatment, 3 times per week for 2 weeks
  Interventions: Device: Sham RAVANS

INTERVENTIONS:
Device: respiratory-gated auricular vagal afferent nerve stimulation (RAVANS) — non-painful electrical stimulation of the auricle
  Other Names: transcutaneous vagus nerve stimulation
  Arms: RAVANS
Device: Sham RAVANS — sham stimulation
  Arms: Sham stimulation

SUMMARY:
This study is to assess if respiratory-gated auricular vagal nerve stimulation (RAVANS) can improve symptoms of post-treatment Lyme disease syndrome

DETAILED DESCRIPTION:
Lyme disease is caused by the tick-borne spirochete bacteria Borrelia burgdoferi and is the most common vector borne illness in the US. A subset of individuals with confirmed Lyme disease go on to experience persistent fatigue, pain, and/or neurocognitive difficulties after treatment that are of sufficient severity to impact quality of life and physical functioning. This chronic condition has since been termed post-treatment Lyme disease syndrome (PTLDS). The cause of PTLDS is not known and currently there are no recommended treatments.

We have hypothesized that some cases of PTLDS may be caused by an infection or inflammatory process on or near the neuroimmune vagus nerve, which communicates the detection of peripheral inflammation to the central nervous system and triggers the sickness response circuitry.

Increasing evidence shows that transcutaneous auricular nerve stimulation (taVNS) can significantly reduce multiple symptoms of stress disorder including depression, cognitive impairment, psychomotor retardation, sleep disturbance. Respiratory-gated auricular vagal afferent nerve stimulation(RAVANS), a type of taVNS, which synchronizes stimulation to the respiratory cycle, modulate vagal systems and optimize stimulations and has been shown beneficial effect in pain management.

In this study, we will conduct a randomized, double blinded, sham-controlled pilot study to explore the effect of RAVANS on the symptoms in individuals diagnosed with PTLDS using psychometric measurement, function and cognitive test, and serum biomarkers.

ELIGIBILITY:
Inclusion Criteria:

1. Adults of all genders ≥ 18 years
2. History of Lyme disease treated with antibiotics, and current PTLDS diagnosed by a physician
3. Evidence of past B. burgdorferi infection based on positive results from both enzyme immunoassay and Western blot testing.
4. Ability to provide informed consent,
5. willing to maintain current PTLDS treatment regimen during participation in the study (if on long-term antibiotics or supplements for PTLDS management).

Exclusion Criteria:

1. History of other neurological disorder that in the judgement of the investigator could interfere with the treatment or the interpretation of the results (e.g., epilepsy, history of stroke, tumor, brain tissue damaging pathologies etc.).
2. Current psychotic disorder (e.g., schizophrenia).
3. Current acute illness or infection (e.g. cold or flu).
4. Current or past history of psychiatric illness; PTSD, depression and anxiety are exclusion criteria only if the conditions are so severe as to have required hospitalization in the past 5 years.
5. History of recurrent vaso-vagal syncope
6. Bradycardia defined as resting heart rate <50bpm
7. Implanted electronic device (e.g., pacemaker, neurostimulator)
8. Use of immunosuppressive medication such as prednisone, TNF medications within 2 weeks of the visit or anticipated use during the study.
9. Current use of anti-inflammatory steroid use.
10. Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2022-05-31 (Actual); Primary Completion 2024-08-11 (Actual); Study Completion 2025-04-25 (Actual)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aranow C, Atish-Fregoso Y, Lesser M, Mackay M, Anderson E, Chavan S, Zanos TP, Datta-Chaudhuri T, Bouton C, Tracey KJ, Diamond B. Transcutaneous auricular vagus nerve stimulation reduces pain and fatigue in patients with systemic lupus erythematosus: a randomised, double-blind, sham-controlled pilot trial. Ann Rheum Dis. 2021 Feb;80(2):203-208. doi: 10.1136/annrheumdis-2020-217872. Epub 2020 Nov 3. PMID 33144299
- [Background] Dantzer R, Konsman JP, Bluthe RM, Kelley KW. Neural and humoral pathways of communication from the immune system to the brain: parallel or convergent? Auton Neurosci. 2000 Dec 20;85(1-3):60-5. doi: 10.1016/S1566-0702(00)00220-4. PMID 11189027
- [Background] Ek M, Kurosawa M, Lundeberg T, Ericsson A. Activation of vagal afferents after intravenous injection of interleukin-1beta: role of endogenous prostaglandins. J Neurosci. 1998 Nov 15;18(22):9471-9. doi: 10.1523/JNEUROSCI.18-22-09471.1998. PMID 9801384
- [Background] Embers ME, Hasenkampf NR, Jacobs MB, Tardo AC, Doyle-Meyers LA, Philipp MT, Hodzic E. Variable manifestations, diverse seroreactivity and post-treatment persistence in non-human primates exposed to Borrelia burgdorferi by tick feeding. PLoS One. 2017 Dec 13;12(12):e0189071. doi: 10.1371/journal.pone.0189071. eCollection 2017. PMID 29236732
- [Background] Garcia RG, Lin RL, Lee J, Kim J, Barbieri R, Sclocco R, Wasan AD, Edwards RR, Rosen BR, Hadjikhani N, Napadow V. Modulation of brainstem activity and connectivity by respiratory-gated auricular vagal afferent nerve stimulation in migraine patients. Pain. 2017 Aug;158(8):1461-1472. doi: 10.1097/j.pain.0000000000000930. PMID 28541256
- [Background] Kong J, Fang J, Park J, Li S, Rong P. Treating Depression with Transcutaneous Auricular Vagus Nerve Stimulation: State of the Art and Future Perspectives. Front Psychiatry. 2018 Feb 5;9:20. doi: 10.3389/fpsyt.2018.00020. eCollection 2018. PMID 29459836
- [Background] Napadow V, Edwards RR, Cahalan CM, Mensing G, Greenbaum S, Valovska A, Li A, Kim J, Maeda Y, Park K, Wasan AD. Evoked pain analgesia in chronic pelvic pain patients using respiratory-gated auricular vagal afferent nerve stimulation. Pain Med. 2012 Jun;13(6):777-89. doi: 10.1111/j.1526-4637.2012.01385.x. Epub 2012 May 8. PMID 22568773
- [Background] VanElzakker MB. Chronic fatigue syndrome from vagus nerve infection: a psychoneuroimmunological hypothesis. Med Hypotheses. 2013 Sep;81(3):414-23. doi: 10.1016/j.mehy.2013.05.034. Epub 2013 Jun 19. PMID 23790471
- [Background] Zubcevik N, Mao C, Wang QM, Bose EL, Octavien RN, Crandell D, Wood LJ. Symptom Clusters and Functional Impairment in Individuals Treated for Lyme Borreliosis. Front Med (Lausanne). 2020 Aug 21;7:464. doi: 10.3389/fmed.2020.00464. eCollection 2020. PMID 32974369

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | RAVANS | Sham Stimulation
Started | 8 | 7
Completed | 8 | 7
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | RAVANS | Sham Stimulation | Total
Number analyzed (Participants) | 8 | 7 | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 5 | 11
  >=65 years | 2 | 2 | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.3 (18.1) | 59.1 (12.6) | 54.4 (15.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 7 | 15
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 8 | 7 | 15
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 8 | 7 | 15
Functional Comorbidity Index [Mean (Standard Deviation); unit: units on a scale] — The Functional Comorbidity Index (FCI) is a tool developed to predict physical function in adults based on their pre-existing chronic health conditions. The FCI is an unweighted, self-reported index of 18 specific chronic conditions. Each condition is scored on a binary scale with 1 point given for the presence of a condition and 0 for the absence. The sum of the individual condition scores yields FCU score; range, 0 to 18. A score of 0 indicates no comorbidities, while a score of 18 indicates the highest burden of comorbid conditions related to physical function.
  units on a scale | 15.1 (1.21) | 14.6 (2.4) | 14.8 (1.9)

OUTCOME MEASURES:

1. Primary Outcome: Horowitz Lyme-Multiple Systemic Infectious Disease Syndrome Questionnaire
Description: This 55-item questionnaire evaluates the frequency, severity, and incidence of Lyme symptoms as well as assessing one's perceived overall health.
  Minimum value:0 Maximum value: 114 The higher number indicates more symptoms
Time Frame: Before treatment (baseline) and Post treatment ( at the end of 2-week treatment)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | RAVANS | Sham Stimulation
Number analyzed (Participants) | 8 | 7
score on a scale
  Before Treatment | 50.5 (21.3) | 44.8 (14.1)
  Post Treatment | 33.8 (17.3) | 25.6 (9.9)
Statistical Analysis 1: Comparison: RAVANS vs Sham Stimulation; Test type: Superiority; p = 0.07, ANOVA
Statistical Analysis 2: Comparison: RAVANS; Test type: Superiority; p = 0.039, t-test, 2 sided
Statistical Analysis 3: Comparison: Sham Stimulation; Test type: Superiority; p = 0.037, t-test, 2 sided

2. Secondary Outcome: Sedentary Behaviors Questionnaire
Description: This 18-item questionnaire asks about the amount of time spent engaged in sedentary behaviors on typical weekdays and weekends.
  Minimum:0 Maximum:162 The higher scores mean higher sedentary behaviors
Time Frame: Before treatment (baseline) and Post treatment (at the end of 2-week treatment)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | RAVANS | Sham Stimulation
Number analyzed (Participants) | 8 | 7
score on a scale
  Before Treatment | 55.8 (11.5) | 49.5 (8.4)
  Post Treatment | 48.8 (22.5) | 52.6 (12.4)
Statistical Analysis 1: Comparison: RAVANS vs Sham Stimulation; Test type: Superiority; p = 0.38, ANOVA
Statistical Analysis 2: Comparison: RAVANS; Test type: Superiority; p = 0.79, t-test, 2 sided
Statistical Analysis 3: Comparison: Sham Stimulation; Test type: Superiority; p = 0.069, t-test, 2 sided

3. Secondary Outcome: Fatigue Symptom Inventory
Description: This non-diagnosis-specific questionnaire measures the severity of fatigue symptoms and how much these factors interfere with the subjects' lives.
  Minimum value:0 Maximum value:127 The higher scores mean higher fatigue symptoms
Time Frame: Before treatment (baseline) and Post treatment (at the end of 2-week treatment)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | RAVANS | Sham Stimulation
Number analyzed (Participants) | 8 | 7
score on a scale
  Before Treatment | 89.4 (20.6) | 65.4 (34.3)
  Post Treatment | 66.8 (31.4) | 44.3 (22.9)
Statistical Analysis 1: Comparison: RAVANS vs Sham Stimulation; Test type: Superiority; p = 0.92, ANOVA
Statistical Analysis 2: Comparison: RAVANS; Test type: Superiority; p = 0.053, t-test, 2 sided
Statistical Analysis 3: Comparison: Sham Stimulation; Test type: Superiority; p = 0.069, t-test, 2 sided

4. Secondary Outcome: Brief Pain Inventory-Pain 24 Hours
Description: This 15-item questionnaire assesses the location, severity, and type of current pain, using analogue scales and body diagrams. Subscale-pain 24 hours describes the pain at its worst in the past 24 hours.
  Minimum value:0 Maximum value: 10 The higher scores means higher pain level
Time Frame: Before treatment (baseline) and Post treatment (at the end of 2-week treatment)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | RAVANS | Sham Stimulation
Number analyzed (Participants) | 8 | 7
score on a scale
  Before Treatment | 5.6 (2.1) | 6.4 (2.2)
  Post Treatment | 4.8 (3.3) | 4.4 (2.9)
Statistical Analysis 1: Comparison: RAVANS vs Sham Stimulation; Test type: Superiority; p = 0.35, ANOVA
Statistical Analysis 2: Comparison: RAVANS; Test type: Superiority; p = 0.59, t-test, 2 sided
Statistical Analysis 3: Comparison: Sham Stimulation; Test type: Superiority; p = 0.073, t-test, 2 sided

5. Secondary Outcome: Beck Depression Inventory
Description: This questionnaire evaluates current depressive symptoms. Minimum value: 0 Maximum value: 63 The higher scores mean higher depressive symptoms
Time Frame: Before treatment (baseline) and Post treatment (at the end of 2-week treatment)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | RAVANS | Sham Stimulation
Number analyzed (Participants) | 8 | 7
score on a scale
  Before Treatment | 42.1 (12.9) | 33.3 (10.9)
  Post Treatment | 33.7 (14.6) | 28 (4.9)
Statistical Analysis 1: Comparison: RAVANS vs Sham Stimulation; Test type: Superiority; p = 0.93, ANOVA
Statistical Analysis 2: Comparison: RAVANS; Test type: Superiority; p = 0.02, t-test, 2 sided
Statistical Analysis 3: Comparison: Sham Stimulation; Test type: Superiority; p = 0.17, t-test, 2 sided

6. Secondary Outcome: Beck Anxiety Inventory
Description: This questionnaire evaluates current anxiety symptoms. Minimum value: 0 Maximum value: 63 The higher scores mean higher anxiety symptoms
Time Frame: Before treatment (at baseline) and after treatment (at the end of 2-week treatment)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | RAVANS | Sham Stimulation
Number analyzed (Participants) | 8 | 7
score on a scale
  Before Treatment | 19.5 (11.1) | 13.1 (0.8)
  Post Treatment | 11.5 (9.9) | 9.3 (6.2)
Statistical Analysis 1: Comparison: RAVANS vs Sham Stimulation; Test type: Superiority; p = 0.29, ANOVA
Statistical Analysis 2: Comparison: RAVANS; Test type: Superiority; p = 0.038, t-test, 2 sided
Statistical Analysis 3: Comparison: Sham Stimulation; Test type: Superiority; p = 0.08, t-test, 2 sided

7. Secondary Outcome: Pittsburgh Sleep Quality Index
Description: This 9-item questionnaire assesses sleep quality and patterns of sleep. Minimum value: 0 Maximum value: 21 The higher scores mean poorer sleep quality
Time Frame: Before treatment (baseline) and Post treatment (at the end of 2-week treatment)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | RAVANS | Sham Stimulation
Number analyzed (Participants) | 8 | 7
score on a scale
  Before Treatment | 13.8 (4.2) | 9.0 (4.2)
  Post Treatment | 9.8 (5.7) | 8.0 (3.9)
Statistical Analysis 1: Comparison: RAVANS vs Sham Stimulation; Test type: Superiority; p = 0.04, ANOVA
Statistical Analysis 2: Comparison: RAVANS; Test type: Superiority; p = 0.007, t-test, 2 sided
Statistical Analysis 3: Comparison: Sham Stimulation; Test type: Superiority; p = 0.15, t-test, 2 sided

8. Secondary Outcome: Timed Up and Go
Description: Measures the time it takes for a person to stand up from a chair, walk 3 meter, turn, walk back, and sit down again.
Time Frame: Before treatment ( baseline) and Post treatment (at the end of 2-week treatment)
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | RAVANS | Sham Stimulation
Number analyzed (Participants) | 8 | 7
seconds
  Before Treatment | 10.5 (3.5) | 9.3 (2.4)
  Post Treatment | 9.5 (2.8) | 8.6 (1.7)

9. Secondary Outcome: Time to Complete 4 Meters at Usual Walking Speed,
Description: Measure usual walk speed
Time Frame: Before treatment (baseline) and Post treatment (at the end of 2-week treatment)
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | RAVANS | Sham Stimulation
Number analyzed (Participants) | 8 | 7
seconds
  Before Treatment | 4.9 (1.1) | 4.6 (0.6)
  Post Treatment | 4.2 (0.9) | 4.3 (1.0)

10. Secondary Outcome: NIH Toolbox Cognition Battery (NIHTB-CB)
Description: The following cognitive domains are assessed: executive function (Flanker inhibitory control and attention); cognitive flexibility (Dimensional Change Card Sort); working memory (List Sorting); short-term memory (Picture Sequence), processing speed (Pattern Comparison), Picture vocabulary and Oral Reading Recognition Tests. An overall composite score that combines these outcomes (Total Cognition Composite Score) is reported here.
  The higher value means better cognitive function. A score at or near 100 indicates ability that is average compared with others nationally. Scores around 115 suggest above-average cognitive ability, while scores around 130 suggest superior ability (in the top 2 percent nationally, based on Toolbox normative data). Conversely, a score around 85 suggests below-average cognitive ability, and a score in the range of 70 or below suggests significant impairment.
Time Frame: Before treatment (at baseline) and Post treatment (at the end of 2-week treatment)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | RAVANS | Sham Stimulation
Number analyzed (Participants) | 8 | 7
score on a scale
  Before Treatment | 109.8 (7.6) | 107.2 (4.7)
  Post Treatment | 118.7 (9.2) | 113.6 (9.1)
Statistical Analysis 1: Comparison: RAVANS vs Sham Stimulation; Test type: Superiority; p = 0.42, ANOVA
Statistical Analysis 2: Comparison: RAVANS; Test type: Superiority; p = 0.001, t-test, 2 sided
Statistical Analysis 3: Comparison: Sham Stimulation; Test type: Superiority; p = 0.06, t-test, 2 sided

11. Secondary Outcome: Serum Level of Inflammatory Cytokines-IL6
Description: To determine if RAVANS treatment affects the level of inflammation
Time Frame: Before treatment (baseline) and Post treatment (at the end of 2-week treatment)
Measure: Mean (Standard Deviation); unit: fg/ml
Arm/Group | RAVANS | Sham Stimulation
Number analyzed (Participants) | 8 | 7
fg/ml
  Before Treatment | 1897 (1658) | 2648 (1920)
  Post Treatment | 2798 (2391) | 2044 (661)

12. Secondary Outcome: Serum Level of Inflammatory Cytokines-IL10
Description: To determine if RAVANS treatment affects the level of inflammation
Time Frame: Before treatment (at baseline) and after treatment (at the end of 2-week treatment)
Measure: Mean (Standard Deviation); unit: fg/ml
Arm/Group | RAVANS | Sham Stimulation
Number analyzed (Participants) | 8 | 7
fg/ml
  Before Treatment | 668 (293) | 742 (308)
  Post Treatment | 616 (159) | 713 (217)

13. Secondary Outcome: Serum Level of Inflammatory Cytokines-TNF Alfa
Description: To determine if RAVANS treatment affects the level of inflammation
Time Frame: Before treatment (baseline) and Post treatment (at the end of 2-week treatment)
Measure: Mean (Standard Deviation); unit: fg/ml
Arm/Group | RAVANS | Sham Stimulation
Number analyzed (Participants) | 8 | 7
fg/ml
  Before Treatment | 473 (95) | 492 (137)
  Post Treatment | 485 (107) | 470 (135)

ADVERSE EVENTS:
Time Frame: within the study period-2 weeks
Arm/Group | RAVANS | Sham Stimulation
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/7
Other Adverse Events (participants affected / at risk) | 3/8 | 1/7
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RAVANS (N=8) | Sham Stimulation (N=7)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) — nausea during stimulation
Dizziness (General disorders) | 1 (1) | 0 (0) — mild dizziness during treatment
Headache (General disorders) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-11-29): https://cdn.clinicaltrials.gov/large-docs/87/NCT04938687/Prot_SAP_000.pdf